CLINICAL TRIAL: NCT03164265
Title: Safety and Preliminary Efficacy of Donor-derived Regulatory Dendritic Cell (DCreg) Infusion and Immunosuppression Withdrawal in Living Donor Liver Transplantation
Brief Title: DCreg in Living Donor Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Angus W. Thomson PhD DSc (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Angus W. Thomson PhD DSc, Distinguished Professor of Surgery and Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY19020267; IND#17271 (Other: FDA)
Record Dates: First submitted 2017-05-10; First posted 2017-05-23 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Living Donor Liver Transplantation
Keywords: Regulatory Dendritic Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Living donor liver transplant recipients receiving donor-derived DCreg infusion. This is a single arm study
  Interventions: Biological: Regulatory Donor-Derived Dendritic Cell infusion

INTERVENTIONS:
Biological: Regulatory Donor-Derived Dendritic Cell infusion — Regulatory dendritic cells that were prepared from a donor leukapheresis will be infused into liver transplant recipients 7 days prior to surgery
  Other Names: DCreg

SUMMARY:
Phase I/II, single center, prospective, open-label, non-controlled, non-randomized, interventional, cohort study in which low risk living donor liver transplant (LDLT) recipients will receive a single infusion of donor-derived DCreg 1 week prior to transplantation. All patients will be maintained on MPA and Tacrolimus (Tac) for the 1st 6 months after transplantation. At that time point, recipients meeting specific criteria will be slowly weaned off MPA per standard of care over a period of 6 months. Participants will then be evaluated for TAC weaning at 1 yr after transplantation. Those who meet specific criteria be weaned off Tac over 6 months . Successfully weaned participants who remain rejection-free will undergo 3 years of follow-up after the last dose of immunosuppression.

DETAILED DESCRIPTION:
Phase I/II, single center, prospective, open-label, non-controlled, non-randomized, interventional, cohort study in which low risk living donor liver transplant (LDLT) recipients will receive a single infusion of donor-derived DCreg with concurrent mycophenolic acid (MPA) therapy (1/2 dose) 1 week prior to transplantation. All patients will be maintained on MPA and Tacrolimus (Tac) for the 1st 6 months after transplantation. At that time point, recipients meeting specific criteria (no rejection and permissive liver function tests (LFTs)) will be slowly weaned off MPA per standard of care over a period of 6 months. Participants will then be evaluated for TAC weaning at 1 yr after transplantation. Those who meet the criteria of no rejection and permissive LFTs will undergo a protocol liver biopsy and proceed to Tac weaning over 6 months if liver biopsy is permissive. Successfully weaned participants who remain rejection-free will undergo 3 years of follow-up after the last dose of immunosuppression. They will undergo a liver biopsy at 1 yr and 3 yrs after immunosuppression withdrawal. Participants who are removed from the study protocol at any time will return to standard of care but will continue to be followed by the study team and may undergo a liver biopsy at the end of the study (4.5 yrs after transplantation). For subjects who return to standard of care (on immunosuppression at end of study), the year 4.5 biopsy will be optional.

ELIGIBILITY:
Inclusion Criteria:

Donors

1. Able to understand and provide informed consent;
2. Male or female between the ages of 18-55;
3. Meet all standard institutional and UNOS criteria for liver donation;
4. For females of childbearing potential, a negative urine or serum pregnancy test;
5. Negative for HIV (5th generation Test and NAT), HTLV-1, HTLV-2;(*)
6. Negative for hepatitis C (antibody and NAT), hepatitis B (surface antigen and NAT)(*)

Recipients

1. Low risk recipient approved for LDLT, irrespective of gender, race, or ethnic background. Low risk is defined by absence of exclusion criteria (below).
2. Between ages 18 and 75 years
3. Undergoing de novo (first) liver transplant
4. Female subjects of childbearing potential must have a negative pregnancy test upon study entry.
5. Agreement to use contraception; according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used from the time that study treatment begins until 1 year after completion of immunosuppression withdrawal.

(*)does not preclude donors from undergoing leukapheresis but cells may not be infused into recipient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Humar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Prospectively enrolled living donor liver transplant recipients pre-op.
Period: Overall Study
Arm/Group | Study Group
Started | 16
Completed | 13
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: 1. subject was excluded from the analysis due to an incidental finding of mucinous adenocarcinoma at the time of transplant.
  2. nd subject experienced a spontaneous pontine hemorrhage 14 days after transplantation with poor prognosis and was withdrawn.
Arm/Group | Study Group
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Safety Events
Description: 1. Safety: Safety will be determined by assessing the percentage of subjects experiencing the following events: i) CTCAE Grade 4 or higher infusion reaction; ii) CTCAE Grade 4 or higher infection; iii) Malignancy other than non-melanoma skin cancer or HCC recurrence; iv) Rejection resulting in recipient death or retransplantation; v) Biopsy-proven severe acute rejection; vi) Any grade chronic rejection; vii) Non-surgical graft loss; viii) Recipient death;
Time Frame: 6 years
Population: living donor liver transplant recipients
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 13
Participants | 1

2. Primary Outcome: Preliminary Efficacy
Description: Proportion of patients able to achieve staged immunosuppression withdrawal with operational tolerance
Time Frame: 2.5 years
Population: living donor liver transplant recipients
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 13
Participants | 3

3. Secondary Outcome: Donor Specific Antigen (DSA) Levels
Description: DSA levels early (<6 weeks) and late (> 6 weeks) after transplantation
Time Frame: 6 years
Population: living donor liver transplant recipients.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 13
Participants
  early DSA | 3
  late DSA | 7
  No DSA | 3

4. Secondary Outcome: Change in Renal Function
Description: Change in renal function measured by change in estimated glomerular filtration rate (eGFR)
Time Frame: from baseline to 4.5 years post transplantation
Population: living donor liver transplant recipients
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Study Group
Number analyzed (Participants) | 13
ml/min | 4.42 (1.5)

5. Secondary Outcome: Change in Quality of Life
Description: Scale title: Short Form 36 (SF-36) Quality of Life questionnaire. Minimum and maximum values 0 to 100 higher scores indicates better health.
Time Frame: 1 year post-transplantation (prior to weaning) 4.5 years post transplantation
Population: living donor liver transplant recipients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm
Number analyzed (Participants) | 13
score on a scale
  Physical functioning | -7.7 (21.82)
  Role limitations due to physical health | -12.5 (29.46)
  Role limitations due to emotional problems | -10 (41.73)
  Energy and fatigue | -3.83 (7.76)
  Emotional well-being | -12.4 (19.64)
  Social functioning | -13.75 (30.31)
  Pain | -13.25 (21.35)
  General health | -11.5 (20.42)
  Health change | -25 (25)

6. Secondary Outcome: Change in Cardiovascular Risk Factors (Systolic Blood Pressure)
Time Frame: from baseline to 4.5 years post transplantation
Population: living donor liver transplant recipients
Measure: Mean (Standard Deviation); unit: millimeters of Mercury (Hg)
Arm/Group | Study Group
Number analyzed (Participants) | 13
millimeters of Mercury (Hg) | 10.5 (16.31)

7. Secondary Outcome: Change in Cardiovascular Risk Factors (Triglycerides)
Time Frame: from baseline to 4.5 years
Population: living donor liver transplant recipients
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Study Group
Number analyzed (Participants) | 13
mg/dL | 98.88 (141.3)

ADVERSE EVENTS:
Time Frame: 4.5 years
Description: same as clinical trials.gov
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=13)
CMV viremia (Infections and infestations) | 2 (2)
Herpes Simplex virus (Infections and infestations) | 1 (1)
COVID infection (Infections and infestations) | 2 (2)
bacterial infection (Infections and infestations) | 3 (3)
oral candidiasis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03164265/Prot_SAP_000.pdf
  • Informed Consent Form: recipient (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03164265/ICF_001.pdf
  • Informed Consent Form: donor (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03164265/ICF_002.pdf